CLINICAL TRIAL: NCT05764785
Title: Evaluating the Acceptability, Feasibility, and Efficacy of a Digital Peer Mentoring Platform With College Student Populations
Brief Title: Evaluating a Digital Peer Mentoring Platform With College Student Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academic Web Pages (Industry)
Collaborators: University of Massachusetts, Boston (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 375649; 1R41MH126795-01A1 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-03-13 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Well-Being, Psychological; Anxiety; Depression; Mentoring to Support the Transition to College
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants assigned based on the timing of their courses in the summer program
Masking Description: Participants will know which condition they are assigned (mentors will know if they are using MentorPRO; students will know if they are using MentorPRO). Researchers will also know participant group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MentorPRO (Experimental): Participants assigned to use MentorPRO
  Interventions: Behavioral: MentorPRO
- Control (No Intervention): Participants in mentoring program as usual

INTERVENTIONS:
Behavioral: MentorPRO — MentorPRO is a novel application and web platform for mentoring programs that allows students to set goals, track their challenges, and find just-in time resources, while connecting to a mentor for personalized support and progress monitoring.
  Arms: MentorPRO

SUMMARY:
The goal of this clinical trial is to test the acceptability, feasibility, and efficacy of MentorPRO, a novel application that connects mentors and mentees, among incoming college first-year students in a public university. The main questions it aims to answer are:

* What is the acceptability and feasibility of the MentorPRO mentoring platform?
* Does mentoring with MentorPRO demonstrate an impact on academic outcomes (i.e., GPA) and indices of wellbeing (i.e., mental health, connectedness, academic self-efficacy, and overall wellbeing) among a diverse sample of incoming or first year college students?

Participants in the MentorPRO group will:

* Use MentorPRO with their assigned mentors to communicate for 9 weeks about transitioning to college and completing a brief summer course at the university
* Complete surveys about their opinions of MentorPRO

All participants (regardless of group assignment) will:

* Complete surveys about their mental health and overall wellbeing
* Work with a mentor throughout participation in a brief summer course at the university

DETAILED DESCRIPTION:
Every student in the identified program this summer (and meets the study eligibility criteria) will be eligible to participate in the study. Students who opt into participation in research activities will complete two brief surveys. Students in the intervention condition will use MentorPRO, which is a novel application and web platform for mentoring programs that allows students to set goals, track their challenges, and find just-in time resources, while connecting to a mentor for personalized support and progress monitoring. All students in in the program will be matched with a peer mentor. Students will be assigned to mentoring using MentorPRO (intervention condition) or as-usual (control condition) based on the timing of their courses; students in the morning courses and virtual courses of the summer program will use MentorPRO. All students involved in the summer program will be involved in one week of orientation, six weeks of academic programming and peer mentoring (June 12th-July 21st), meeting four days per week during the summer prior to mentees' first year in college, as well as two weeks of post-program peer mentoring (total trial of nine weeks).

At the beginning of their membership with the program, all students and mentors will be invited to participate in additional research activities. Recruitment invitations will be in postcard format from Dr. Jean Rhodes or from program staff, explaining what the study is about, what is involved for participants, what the eligibility criteria is, and a link to a Qualtrics form. The Qualtrics link will have (in order): an informed consent, an eligibility screener, and if eligible, and the pre-intervention survey (Time 1; T1). Program leaders will also promote the research project during program time, in which staff will use the same language provided in the recruitment email and flier. Students will also have time to ask questions, and any questions in which program staff cannot answer will be escalated to the research team. Individuals will also be provided the contact information of the study Principal Investigator (Dr. Jean Rhodes) in the consent form so that they can ask any questions before consenting, if relevant.

Student mentees: All interested participants will let us know their age (to determine whether they complete an informed consent or their parent/guardian completes the informed consent), and then will read and sign an informed consent, after having time to ask questions to program staff and the research team. Then, they will complete an eligibility screener, and if eligible will complete the rest of the baseline survey. Interested and eligible participants will then be prompted to take the pre-intervention survey after consenting to the study (T1). All students consenting to participate will be assigned to a peer mentor in the program. Each peer mentor will be assigned to provide mentoring as usual (without MentorPRO) or provide mentoring via MentorPRO. Students will complete the summer course for 6 weeks following a week of orientation, and will receive peer mentoring during that time. For two weeks after the course, students will be able to contact their peer mentor with questions. At the end of the 9-week trial, students will receive a final survey (T2). The eligibility screener, informed consent, and the surveys will be administered via a Qualtrics link. At the conclusion of their participation, all participants will receive a debriefing statement explaining the study and where to find additional resources if needed.

Intervention condition: In addition to the training in program policies and relationship building provided to program peer mentors, mentors in the MentorHub UMB group will undergo training designed by the research team. Mentors will complete a brief (30-min) online videos and orientation to the MentorHub UMB technology, followed by a 30-min interactive online course on providing supportive accountability, through MentorHub UMB Academy which includes "knowledge checks" to ensure mentors are engaged and understanding the material and tracks progress to ensure course completion. Additional courses will be available to mentors through the academy, including a course on mentoring ethics. Following the online training, groups of mentors will engage in a live web-conference (zoom) session with at least one staff member from UMB and at least one member of the research team, who will use motivational interviewing techniques to ensure mentor buy-in and engagement and review content from the online training modules with mentors. Finally, mentees will be given access to an online orientation to MentorHub UMB, which walks them through instructions about how to download and use the app. All study participants (mentors and student mentees) will have access to tech support within 24 hours from Academic Web Pages for any questions or issues that arise.

Mentors in the intervention condition may recommend students to use a third-party mental health app (Healthy Minds Program; HMP) if needed and provide supportive accountability (i.e., encouragement, nudges, etc) to promote consistent active engagement with HMP. Data on students' engagement with HMP will be provided at the end of the trial from the Healthy Minds team (exported from Amazon Web Services by the research team). Mentors will be encouraged provide weekly supportive accountability to students using Healthy Minds.

Mentors: At the end of the summer program, mentors will be recruited to complete a survey. Interested mentors will fill out an eligibility screener, and, if eligible, an informed consent form and brief demographics survey (all through Qualtrics), and survey with asking about their experiences as a mentor.

ELIGIBILITY:
Inclusion criteria:

* Being a current member of the identified summer program (Directions for Student Potential at the University of Massachusetts Boston during the 2023 summer)
* Can speak, read, and write in English
* Has access to a smartphone
* 18-years-old or older
* Any self-reported symptoms of anxiety, depression, life dissatisfaction, or lack of college belonging

Exclusion criteria:

* Not a member of the identified summer program (Directions for Student Potential at the University of Massachusetts Boston during the 2023 summer)
* No access to smartphone
* Cannot speak, read, and write in English
* under 18-years-old
* Not reporting any symptoms of anxiety, depression, life dissatisfaction, or lack of college belonging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean E Rhodes, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were assigned to their conditions at enrollment.
Period: Overall Study
Arm/Group | MentorPRO | Control
Started | 25 | 38
Completed | 23 | 30
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MentorPRO | Control | Total
Number analyzed (Participants) | 25 | 38 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 38 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Although all participants reported that they were at least 18-years-old, one participant did not report exact age.
  years
    number analyzed (Participants) | 25 | 37 | 62
    (all) | 18.36 (.7) | 18.11 (.39) | 18.21 (.55)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 11 | 18 | 29
  Female | 13 | 19 | 32
  Non-binary | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 30
  Not Hispanic or Latino | 10 | 18 | 28
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 1 | 13 | 14
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 25 | 38 | 63
Self-reported depression symptoms [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire - 9 (PHQ-9): Depression symptoms over the last two weeks, minus item 9 (suicidal ideation) Scores range from 0 (no depression symptoms) to 24 (high/extreme depression symptoms).
  units on a scale | 7.28 (5.81) | 5.76 (4.21) | 6.37 (4.92)
Self-reported anxiety symptoms [Mean (Standard Deviation); unit: units on a scale] — General Anxiety Disorder - 7 (GAD-7): Anxiety symptoms over the last two weeks Scores range from 0 (no anxiety symptoms) to 21 (extreme/severe anxiety symptoms)
  units on a scale | 6.36 (5.74) | 4.13 (5.20) | 5.02 (5.48)
Academic self-efficacy [Mean (Standard Deviation); unit: units on a scale] — Single item of feelings of academic self-efficacy: I am confident that I will be a successful student at UMass Boston.
  Scores range from strongly disagree (1) to strongly agree (5) Greater scores reflect greater perceived academic self-efficacy Population: One participant preferred not to respond to this question
  units on a scale
    number analyzed (Participants) | 24 | 38 | 62
    (all) | 4.04 (1.04) | 4.39 (.79) | 4.26 (.9)
Perceived cognitive load [Mean (Standard Deviation); unit: units on a scale] — Single item assessing cognitive load of finding resources on campus: It can be exhausting to find the information and resources I need to succeed.
  Scores range from strongly disagree (1) to strongly agree (5) Greater scores reflect greater perceived exhaustion when finding needed resources
  units on a scale | 2.88 (1.17) | 2.76 (1.00) | 2.81 (1.06)
Life satisfaction [Mean (Standard Deviation); unit: units on a scale] — Single item of current life satisfaction: In general, how satisfied are you with your life? Responses ranging from 1 (very satisfied) to 4 (very dissatisfied) Increases in scores relate to worsening life satisfaction overall Population: One participant preferred not to answer this question
  units on a scale
    number analyzed (Participants) | 24 | 38 | 62
    (all) | 1.83 (.82) | 2.13 (.96) | 2.02 (.91)
Sense of belonging to university [Mean (Standard Deviation); unit: units on a scale] — Single item assessing feelings of sense of belonging: I feel part of the UMass Boston community.
  Scores range from strongly disagree (1) to strongly agree (5) Greater scores reflect greater sense of belonging to the university community
  units on a scale | 3.76 (1.01) | 3.95 (1.09) | 3.87 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Depression Symptoms
Description: Patient Health Questionnaire - 9 (PHQ-9): Depression symptoms over the last two weeks, minus item 9 (suicidal ideation) Scores range from 0 (no depression symptoms) to 24 (high/extreme depression symptoms).
Time Frame: 9 weeks after program start
Population: Some participants opted to skip this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MentorPRO | Control
Number analyzed (Participants) | 23 | 26
score on a scale | 8.21 (4.97) | 3.88 (3.29)
Statistical Analysis 1: Comparison: MentorPRO vs Control; Test type: Superiority; p = .182, Mixed ANOVA — Assumption of Sphericity was violated and Greenhouse-Geisser was above .75, thus Huynh-Feldt correction was used

2. Primary Outcome: Self-reported Anxiety Symptoms
Description: General Anxiety Disorder - 7 (GAD-7): Anxiety symptoms over the last two weeks Scores range from 0 (no anxiety symptoms) to 21 (extreme/severe anxiety symptoms)
Time Frame: 9 weeks after program start
Population: Some participants opted to skip this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MentorPRO | Control
Number analyzed (Participants) | 23 | 26
score on a scale | 6.39 (5.01) | 3.19 (3.89)
Statistical Analysis 1: Comparison: MentorPRO vs Control; Test type: Superiority; p = .461, Mixed ANOVA — Assumption of Sphericity was violated and Greenhouse-Geisser was above .75, thus Huynh-Feldt correction was used

3. Primary Outcome: Life Satisfaction
Description: Single item of current life satisfaction: In general, how satisfied are you with your life? Responses ranging from 1 (very satisfied) to 4 (very dissatisfied)
Time Frame: 9 weeks after program start
Population: Some participants opted to skip this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MentorPRO | Control
Number analyzed (Participants) | 22 | 27
units on a scale | 2.00 (.98) | 1.96 (.94)
Statistical Analysis 1: Comparison: MentorPRO vs Control; Test type: Superiority; p = .228, Mixed ANOVA — Assumption of Sphericity was violated and Greenhouse-Geisser was above .75, thus Huynh-Feldt correction was used

4. Secondary Outcome: Academic Self-efficacy
Description: Single item of feelings of academic self-efficacy: I am confident that I will be a successful student at UMass Boston.
  Scores range from strongly disagree (1) to strongly agree (5) Greater scores reflect greater perceived academic self-efficacy
Time Frame: 9 weeks after program start
Population: Some participants opted to skip this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MentorPRO | Control
Number analyzed (Participants) | 23 | 27
units on a scale | 3.61 (1.27) | 4.41 (.69)
Statistical Analysis 1: Comparison: MentorPRO vs Control; Test type: Superiority; p = .295, Mixed ANOVA — Assumption of Sphericity was violated and Greenhouse-Geisser was above .75, thus Huynh-Feldt correction was used

5. Secondary Outcome: Cognitive Load
Description: Single item assessing cognitive load of finding resources on campus: It can be exhausting to find the information and resources I need to succeed.
  Scores range from strongly disagree (1) to strongly agree (5) Greater scores reflect greater perceived exhaustion when finding needed resources
Time Frame: 9 weeks after program start
Population: Some participants opted to skip this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MentorPRO | Control
Number analyzed (Participants) | 23 | 27
units on a scale | 2.87 (1.22) | 2.74 (1.10)
Statistical Analysis 1: Comparison: MentorPRO vs Control; Test type: Superiority; p = .915, Mixed ANOVA — Assumption of Sphericity was violated and Greenhouse-Geisser was above .75, thus Huynh-Feldt correction was used

6. Secondary Outcome: Sense of Belonging to the University Community
Description: Single item assessing feelings of sense of belonging: I feel part of the UMass Boston community.
  Scores range from strongly disagree (1) to strongly agree (5) Greater scores reflect greater sense of belonging to the university community
Time Frame: 9 weeks after program start
Population: Some participants opted to skip this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MentorPRO | Control
Number analyzed (Participants) | 23 | 27
units on a scale | 3.57 (1.24) | 4.26 (.94)
Statistical Analysis 1: Comparison: MentorPRO vs Control; Test type: Superiority; p = .226, Mixed ANOVA — Assumption of Sphericity was violated and Greenhouse-Geisser was above .75, thus Huynh-Feldt correction was used

ADVERSE EVENTS:
Time Frame: Two months
Arm/Group | MentorPRO | Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/30
Other Adverse Events (participants affected / at risk) | 0/23 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05764785/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05764785/SAP_001.pdf
  • Informed Consent Form (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05764785/ICF_002.pdf